CLINICAL TRIAL: NCT06095089
Title: A Phase 1 Study of JNJ-87189401 (PSMA-CD28 Bispecific Antibody) Combined With JNJ-78278343 (KLK2-CD3 Bispecific Antibody) for Advanced Prostate Cancer
Brief Title: A Study of JNJ-87189401 Plus JNJ-78278343 for Advanced Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR109330; 87189401PCR1001 (Other: Janssen Research & Development, LLC); 2023-504063-17-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2023-10-18; First posted 2023-10-23 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Advanced Prostate Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Part 1 (Dose Escalation) and Part 2 (Dose Expansion) (Experimental): Participants will receive JNJ-78278343+JNJ-87189401 escalated sequentially in Part 1 to select a recommended Phase 2 regimen (RP2R). Participants will receive the combination treatment at the RP2R in Part 2 in different disease settings.
  Interventions: Drug: JNJ-78278343; Drug: JNJ-87189401

INTERVENTIONS:
Drug: JNJ-78278343 — JNJ-78278343 will be administered.
  Other Names: KLK2-CD3; Pasritamig
Drug: JNJ-87189401 — JNJ-87189401 will be administered.
  Other Names: PSMAxCD28

SUMMARY:
The purpose of the study is to determine the recommended regimen for Phase 2 (RP2Rs) of combination of JNJ-87189401 with JNJ-78278343 (Part 1: dose escalation) and further evaluate the safety at RP2Rs (Part 2: dose expansion) in participants with advanced prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate. Adenocarcinoma with small cell or neuroendocrine (NE) features is permitted. However, small cell carcinoma, carcinoid tumor, mixed NE carcinoma, or large cell NE carcinoma is disallowed
* Measurable or evaluable disease per PCWG3 criteria
* Part 1, Part 2A and Part 2B: Prior orchiectomy or medical castration; participants who have not undergone orchiectomy, must be receiving ongoing androgen deprivation therapy with a gonadotropin releasing hormone (GnRH) analog (agonist or antagonist), prior to the first dose of study drug and must continue this therapy throughout the treatment phase
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Active autoimmune disease within the 12 months prior to signing consent that requires systemic immunosuppressive medications (example, chronic corticosteroids, methotrexate, or tacrolimus)
* Any of the following within 6 months prior to signature of informed consent: a. myocardial infarction, b. severe or unstable angina, c. clinically significant ventricular arrhythmias, d. congestive heart failure (New York Heart Association [NYHA] class II to IV), e. transient ischemic attack, and f. Cerebrovascular accident

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 250 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2027-06-21 (Estimated); Study Completion 2027-10-27 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants With Dose Limiting Toxicity (DLT) | Up to 21 days after first combination dose of study drugs
  DLTs are specific adverse events (AEs) and are defined as any of the following: high grade non-hematologic toxicity or hematologic toxicity.
Part 1 and Part 2: Number of Participants with Adverse Events (AEs) by Severity | Up to 3 years 7 months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 with the exception of cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome events, which will be graded by American Society for Transplantation and Cellular Therapy (ASTCT) guidelines. Severity scale ranges from grade 1 (mild) to grade 5 (death). Grade 1= mild, Grade 2= moderate, Grade 3= severe, Grade 4= life-threatening and Grade 5= death related to adverse event.

SECONDARY OUTCOMES:
Part 2: Serum Concentration of JNJ-87189401 | Up to 3 years 7 months
  Serum samples will be analyzed to determine concentrations of JNJ-87189401.
Number of Participants With Antibodies to JNJ-87189401 and JNJ-78278343 | Up to 3 years 7 months
  Number of participants with antibodies to JNJ-87189401 and JNJ-78278343 will be reported.
Objective Response Rate (ORR) | Up to 3 years 7 months
  ORR is defined as the proportion of participants who have a partial response (PR) or better according to response evaluation criteria in solid tumors (RECIST) version 1.1 without evidence of bone progression according to Prostate Cancer Working Group 3 (PCWG3).
Radiographic Progression-Free Survival (rPFS) | Up to 3 years 7 months
  rPFS is defined time from the date of first dose of study drug until the date of objective disease progression or death, whichever comes first.
Prostate Specific Antigen (PSA) Response Rate | Up to 3 years 7 months
  PSA response rate is defined as the percentage of participants with a confirmed decline of PSA of 50 percent (%) or more from baseline.
Duration of Response (DOR) | Up to 3 years 7 months
  DOR is defined for participants who achieved response (PR or better) as the time between the date of initial documentation of response (PR or better) to the date of first documented evidence of progressive disease, as defined in the PCWG3, or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (5):
- United States (3):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Herbert Irving Comprehensive Cancer Center Columbia University Medical Center, New York, New York
  - South Texas Accelerated Research Therapeutics, LLC (START), San Antonio, Texas
- France (2):
  - Centre Leon Berard, Lyon
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency